CLINICAL TRIAL: NCT01411397
Title: Mesh Hernioplasty Of Strangulated Hernias With Intestinal Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: mansoura university, mansoura university
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: strangulated hernia
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2005-06

CONDITIONS: Strangulated Hernia
Keywords: Infection; Prosthesis; Recurrence; Strangulation
MeSH Terms: conditions — Infections; Recurrence | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesh repair (Active Comparator): MESH HERNIA REPAIR WHEN REqUIRE INTESTINAL RESECTION
  Interventions: Other: SURGERY
- mesh repair without intestinal resection (Active Comparator): mesh repair of strangulated hernia without resection
  Interventions: Other: mesh repair

INTERVENTIONS:
Other: SURGERY — REPAIR OF STRANGULATED HERNIA with intestinal resection
  Other Names: mesh hernioplasty
  Arms: mesh repair
Other: mesh repair — mesh repair of strangulated hernia without resection
  Other Names: mesh hernioplasty without resection
  Arms: mesh repair without intestinal resection

SUMMARY:
Primary suture repair increases the risk for recurrence, the fact of benefit of mesh repair in elective situations is documented, and many studies have reported beneficial outcomes of mesh hernioplasty in emergency situations. Still there is controversy of using such grafts in presence of intestinal resection.

DETAILED DESCRIPTION:
Patients with acutely incarcerated hernias (with small intestine contents) who underwent polypropylene mesh hernioplasty were included in this prospective study from June 2005 through Jan. 2011, patients were categorized into 2 groups who required intestinal resection anastomosis (group I)or not (group II).

ELIGIBILITY:
Inclusion Criteria:

* strangulated hernias

Exclusion Criteria:

* above 75, under 18
* recurrent hernia
* peritonitis
* pure omentum contents ASA above 3

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2005-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
wound infection | 5 weeks

SECONDARY OUTCOMES:
operative time | 3hours
  the time from skin incision up to skin closure
morbidity | 5 months
  the perioperative complications
recurrence of the hernia | 6months
  Recurrence of the hernia was defined as an apparent swelling or a palpable defect at the previous surgery site detected clinically or radiologically by ultrasound if needed

CONTACTS AND LOCATIONS:
Overall Officials: ramadan ellithy, md, Study Director — Mansoura University
Locations (1):
- Mohamed Abdellatif, Al Mansurah, Mansoura, Egypt